CLINICAL TRIAL: NCT00662766
Title: Intervention Study on the Health Beneficial Effects of Bread Enriched With Black Currant Seed Press Residues in Healthy Subjects
Brief Title: Intervention With Black Currant Seed Press Residues in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Dr. G. Jahreis, Universitiy of Jena
Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: LSEP H22-05
Record Dates: First submitted 2008-04-10; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Smoking
Keywords: Black currant; Berry seed; Press residue; Tocopherol; Fatty acids; Fiber; Total phenols; TEAC; Comet assay; Dihydroxybenzoic acid
MeSH Terms: conditions — Smoking | interventions — Bread

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: black currant seed press residue — Black currant seed press residue, baked into bread
Dietary Supplement: Bread without black currant seed press residues — Same bread but without seeds
Dietary Supplement: Baseline data — No supplement was administered.

SUMMARY:
The study was performed to investigate the effects of the consumption of black currant seed press residues, which were baked into bread.

DETAILED DESCRIPTION:
Berry seeds are a by-product of berry fabrication (e. g. to juices or jam). In order to maintain their functionality and long life span, berry seeds need to contain cell stabilizing ingredients such as vitamins and polyphenols. Since it seems to be a valuable source of health beneficial substances in human nutrition, commercial use should be found. Therefore, seeds were pressed (seed press residue), ground and baked into bread for consumption.

Black currant seed press residues are rich in tocopherols and also contain anthocyanins; both act as antioxidants. Additionally there is 50% fibre in the residue, soluble and insoluble fibre in equal shares.

ELIGIBILITY:
Inclusion Criteria:

* discrimination between smoker (> 5 cigarets/d) or non-smoker

Exclusion Criteria:

* diet during the study
* serious sport
* diagnosed diseases
* use of nutritional supplements

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
oxidant/antioxidant status of the test person | after 1, 5, and 9 weeks

SECONDARY OUTCOMES:
tocopherol intake, tocopherol faecal excretion and serum tocopherol concentration | after 1, 5, and 9 weeks
fiber intake and excretion | after 1, 5, and 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Study Chair — University of Jena, Dept. of Nutritional Physiology; Dorit Helbig, Dipl. troph., Principal Investigator — University of Jena, Dept. of Nutritional Physiology

REFERENCES:
- [Derived] Helbig D, Wagner A, Schubert R, Jahreis G. Tocopherol isomer pattern in serum and stool of human following consumption of black currant seed press residue administered in whole grain bread. Clin Nutr. 2009 Dec;28(6):662-7. doi: 10.1016/j.clnu.2009.05.003. Epub 2009 Jun 11. PMID 19523725